CLINICAL TRIAL: NCT03710980
Title: Accuracy of Pulse Oximeters With Profound Hypoxia
Status: Completed | Type: Observational
Sponsor: Hancock Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: BEDD01
Record Dates: First submitted 2018-10-16; First posted 2018-10-18 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Oximetry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Healthy Adult Volunteer
  Interventions: Device: Oximeter

INTERVENTIONS:
Device: Oximeter — Participants breathe a controlled gas mixture to induce several reduced oxygen states while oximeter measurements are taken for comparison to corresponding arterial blood draw samples to assess oximeter accuracy.

SUMMARY:
This study to assess the oxygen saturation accuracy of the Beddr SleepTuner in profound hypoxia.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is male or female, aged ≥18 and <50.
2. The subject is in good general health with no evidence of any medical problems.
3. The subject is fluent in both written and spoken English.
4. The subject has provided informed consent and is willing to comply with the study procedures.

Exclusion Criteria:

1. The subject is obese (BMI>30).
2. The subject has a known history of heart disease, lung disease, kidney or liver disease.
3. Diagnosis of asthma, sleep apnea, or use of CPAP.
4. Subject has diabetes.
5. Subject has a clotting disorder.
6. The subject a hemoglobinopathy or history of anemia, per subject report or the first bloodsample, that in the opinion of the investigator, would make them unsuitable for study participation.
7. The subject has any other serious systemic illness.
8. The subject is a current smoker.
9. Any injury, deformity, or abnormality at the sensor sites that in the opinion of the investigators' would interfere with the sensors working correctly.
10. The subject has a history of fainting or vasovagal response.
11. The subject has a history of sensitivity to local anesthesia.
12. The subject has a diagnosis of Raynaud's disease.
13. The subject has unacceptable collateral circulation based on exam by the investigator (Allen's test).
14. The subject is pregnant, lactating or trying to get pregnant.
15. The subject is unable or unwilling to provide informed consent, or is unable or unwilling to comply with study procedures.
16. The subject has any other condition, which in the opinion of the investigators' would make them unsuitable for the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adult volunteers.
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2018-09-19 (Actual); Study Completion 2018-09-19 (Actual)

PRIMARY OUTCOMES:
SpO2 Accuracy | 60 minutes
  Collect and analyze data to determine SpO2 accuracy of oximeters under test.

CONTACTS AND LOCATIONS:
Locations (1):
- UCSF Hypoxia Lab, San Francisco, California, United States